CLINICAL TRIAL: NCT03640702
Title: The Effect of Primary Cesarean Section Prevention on Maternal and Neonatal Outcomes
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Kamel Mattar MD, Principal Investigator, Rambam Health Care Campus
Other Study IDs: 0258-17-RMB
Record Dates: First submitted 2018-08-14; First posted 2018-08-21 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Cesarean Section Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prolonged second stage of labor: Women with prolonged second stage of labor as specified before.
  Interventions: Other: Protocol change

INTERVENTIONS:
Other: Protocol change — To examine the effect of prolonging the second stage of labor on the rate of cesarean delivery, maternal and neonatal outcomes

SUMMARY:
The study aimed to examine the effect of prolonging the second stage of labor on the rate of Cesarean section (CS), maternal and neonatal outcomes.

The study compared 2 time periods. The first time period was between May 2011 until April 2014 when a prolonged second stage in nulliparous women was considered three hours with regional anesthesia or two hours if no such anesthesia was provided. Second stage arrest was defined in multiparous women after two hours with regional anesthesia or one hour without it. The second time period was between May 2014 until April 2017, allowed nulliparous and multiparous women to continue the second stage of labor an additional one hour before diagnosing second-stage arrest. Singleton deliveries at or beyond 37 weeks' gestation were initially considered for eligibility.

DETAILED DESCRIPTION:
The study aimed to examine the effect of prolonging the second stage of labor on the rate of Cesarean section (CS), maternal and neonatal outcomes.

The study compared 2 time periods. The first time period was between May 2011 until April 2014 when a prolonged second stage in nulliparous women was considered three hours with regional anesthesia or two hours if no such anesthesia was provided. Second stage arrest was defined in multiparous women after two hours with regional anesthesia or one hour without it. The second time period was between May 2014 until April 2017, allowed nulliparous and multiparous women to continue the second stage of labor an additional one hour before diagnosing second-stage arrest. Singleton deliveries at or beyond 37 weeks' gestation were initially considered for eligibility.

The rate of CS, operative vaginal deliveries, 3rd and 4th degree lacerations, postpartum hemorrhage, arterial cord PH below 7 and admissions to the neonatal intensive care unit (NICU).

ELIGIBILITY:
Inclusion Criteria:

1. Singleton deliveries at or beyond 37 weeks' gestation.

Exclusion Criteria:

1. Non-vertex presentation.
2. Trial of labor after CS.
3. High risk pregnancy (multiple gestation, preeclampsia, diabetes mellitus, intrauterine growth restriction).
4. Known fetal anomalies and intrauterine fetal demise.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female
Study Population: Pregnant women in labor
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
The rate of primary CS. | Between 2011 and 2017.
  The rate of primary CS in percentage of the total participants.

SECONDARY OUTCOMES:
The rate of operative vaginal delivery. | Between 2011 and 2017.
  The rate of operative vaginal delivery in percentage of the total participants.
Post-partum hemorrhage. | Between 2011 and 2017.
  Post-partum hemorrhage as estimated in liters.
The need for blood transfusion. | Between 2011 and 2017.
  Number and type of blood products required post-partum and calculation of the number of patients that required blood products out of the total number of participants in percentage.
Third-and fourth-degree laceration rate. | Between 2011 and 2017.
  Third-and fourth-degree laceration rate of the total number of participants.
Chorioamnionitis rate. | Between 2011 and 2017.
  Chorioamnionitis rate in percentage of the total participants.
Admission to the NICU. | Between 2011 and 2017.
  Admission to the NICU in percentage of the total participants.

CONTACTS AND LOCATIONS:
Overall Officials: Kamel Mattar, MD, Principal Investigator — Principal Investigator
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No